CLINICAL TRIAL: NCT03626116
Title: What Determines Satisfaction of Patients With Rheumatoid Arthritis After Hand Reconstruction Using Silicone Metacarpophalangeal Arthroplasty
Brief Title: Patient Satisfaction After Silicone Metacarpophalangeal Arthroplasty
Status: Completed | Type: Observational
Sponsor: Schulthess Klinik (Other)
Responsible Party: Sponsor
Other Study IDs: MCP Arthroplasty RA patients
Record Dates: First submitted 2018-07-19; First posted 2018-08-10 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Rheumatoid Arthritis - Hand Joint

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: silicone metacarpophalangeal arthroplasty (SMPA) — Replacement of the metacarpophalangeal (MCP) joint using a silicone arthroplasty

SUMMARY:
The primary objective of this study is to identify determinants of long-term patient satisfaction after hand reconstruction using silicone metacarpophalangeal arthroplasty (SMPA). The investigators hypothesize that appearance of the hand, ulnar drift, range of motion, pain, hand function and intake of the newer antirheumatic drugs (i.e. biologicals) influence patient satisfaction.

DETAILED DESCRIPTION:
This is an ambidirectional, monocenter research project consisting of a retrospective chart review and a prospective cohort project.

Participants fulfilling all of the following inclusion criteria are eligible for the project:

* Patients with rheumatoid Arthritis (RA) / Psoriasisarthritis / Lupus erythomatodes who had a SMPA between Jan 2007 and one year before the project examination
* Informed Consent as documented by signature

The presence of any one of the following exclusion criteria will lead to exclusion of the participant:

* Major surgery at another joint at the hand (e.g. proximal interphalangeal (PIP) joint arthroplasty, thumb trapeziectomy) less than 6 months ago
* Legal incompetence
* German language barrier to complete the questionnaires

ELIGIBILITY:
Inclusion Criteria:

* Patients with RA / Psoriasisarthritis / Lupus erythomatodes who had a SMPA between Jan 2007 and one year before the project examination
* Informed Consent as documented by signature

Exclusion Criteria:

* Major surgery at another joint at the hand (e.g. PIP arthroplasty, thumb trapeziectomy) less than 6 months ago
* Legal incompetence
* German language barrier to complete the questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with RA / Psoriasisarthritis / Lupus erythomatodes who had a SMPA
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2018-07-18 (Actual); Primary Completion 2018-12-19 (Actual); Study Completion 2018-12-19 (Actual)

PRIMARY OUTCOMES:
Satisfaction with the treatment result assessed on a 5-point Likert Scale | at least one year after surgery
  The primary outcome is the satisfaction with the treatment result at least one year after surgery and its determinants.
  It will be quantified using this question: How satisfied are you with the overall result of the SMPA surgery? The response options are: Very satisfied (score 1), somewhat satisfied (score 2), neither satisfied nor unsatisfied (score 3), somewhat unsatisfied (score 4), very unsatisfied (score 5).
  For further analyses, this question can be dichotomized into the categories of "satisfied patients" (very satisfied / satisfied) and "unsatisfied patients" (neither satisfied nor dissatisfied or worse).

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Schindele, MD, Principal Investigator — Schulthess Klinik
Locations (1):
- Schulthess Klinik, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No